CLINICAL TRIAL: NCT05850949
Title: The Effect of Konjac Grain in the Post-prandial Glycaemic Response of Healthy Subjects
Acronym: Konjac
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Katolik Widya Mandala Surabaya (Other)
Responsible Party: Principal Investigator, Hendy Wijaya, Head of Clinical Pharmacology research laboratories, Universitas Katolik Widya Mandala Surabaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0015/WM12/KEPK/DSN/T/2023
Record Dates: First submitted 2023-03-29; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Repeated single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Konjac-Grain (Experimental): Without supplementation, followed by Supplementation with Konjac grain from PT. AMBICO
  Interventions: Dietary Supplement: Konjac Grain

INTERVENTIONS:
Dietary Supplement: Konjac Grain — Without supplementation, followed by Supplementation with Dietary Fibre the Konjac-Grain week 1, repeated until week 6, blood collected with a fine needle 10ml citrate-Tube Glucose was measured with disposable 'test-strip', which is then inserted into an electronic blood glucose meter (device: Accu-Check Instant S Glucose from Roche) . Normal value:70 to 99 mg/dL (3.9 to 5.5 mmol/L). Further HbA1c (glycated Hemoglobin A1c) concentration was checked with disposable 'test-strip', which is then inserted into an electronic HbA1c meter (device: Accu-Check Instant S HbA1c from Roche). Unit value fir HbA1c = mg/dl

SUMMARY:
determine the effect of giving the Konjac-Grain formula as a mixture of white rice in suppressing post-prandial glucose absorption.

DETAILED DESCRIPTION:
To determine the effect of giving the Konjac-Grain formula as a mixture of white rice in suppressing post-prandial glucose absorption.

Benefits of research

1. Scientific benefits Add insight into basic science in the field of metabolic physiology and as a scientific reference in the field of nutrition regarding the benefits of konjac grain in helping to improve blood glucose levels.
2. Practical benefits Providing information, education and knowledge to the public that dietary fiber in the form of konyaku grains is a functional food fiber that has the potential to be useful in improving blood glucose levels.

Length of Research Time:

This research will be carried out for approximately 6 weeks and the treatment will be carried out on the first day of each week. The new treatment was repeated the following week.

Notice of Research Results The blood glucose level examination results will be recorded and given to the test subject on the same day or at the next examination.

Research procedure On the first day of every week the patient will be asked to fast at night for 10-12 hours, then the next day, the subjects are given a ready-to-eat meal treatment with rice mixed with the Konjac-Grain grain formula. After eating, blood glucose levels were measured every 30 minutes for 2 hours. This procedure is repeated weekly with different rice: the Konjac-Grain ratio.

The test subject is asked to sign and write down the date on the consent confirmation sheet to participate as a respondent in this study. The test subject's participation in this research is voluntary. The test subject has the full right to withdraw or cancel participation at anytime. All information on the results of your blood tests is confidential.

The test subject's blood will be collected. This procedure will cause pain in the injection area and blood collection. So far there has never been a report that giving the Konjac-Grain grains or other dietary fiber can cause significant health side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, aged 18-50 years
2. Not currently taking any medication
3. Do not have a history of metabolic diseases such as hypertension, prediabetes, metabolic syndrome, non-alcoholic fatty liver disease (NAFLD) previously from the results of doctor and laboratory examinations.
4. Agree to be included as a research subject (by signing an informed consent)

Exclusion Criteria:

1. Was experiencing an acute infectious disease at the time of the study
2. Lack of sleep or heavy physical activity during the study
3. Subjects experienced pregnancy during the study
4. Subjects withdrew at any time during the research

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2023-05-16 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change Post prandial blood glucose | 2 hours after meals.
  Without supplementation, followed by Supplementation with Dietary Fibre the Konjac-Grain week 1, repeated until week 6, blood collected 2 hours after meals with a 3" fine needle 10ml Citrat-Tube
  blood Glucose (mg/dl or mmol/L) one drop (50microliter) of blood from citrat-Tube was transferred to the Glucose test strip. Glucose was measured with disposable 'test-strip', which is then inserted into an electronic blood glucose meter (device: Accu-Check Instant S Glucose from Roche) .
  Normal value:70 to 99 mg/dL (3.9 to 5.5 mmol/L).
Change Post prandial blood HbA1c | 2 hours after meals.
  Without supplementation, followed by Supplementation with Dietary Fibre the Konjac-Grain week 1, repeated until week 6, blood collected 2 hours after meals with a 3" fine needle 10ml Citrat-Tube
  blood HbA1c (mg/dl) one drop (50microliter) of blood from citrat-Tube was transferred to the HbA1c test strip. HbA1c was measured with disposable 'test-strip', which is then inserted into an electronic blood glucose meter (device: Accu-Check Instant S HbA1c from Roche) .
  Normal value:80-180 mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Katolik Widya Mandala Surabaya, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Share after publication